CLINICAL TRIAL: NCT03753009
Title: Iontophoretic Transepithelial Collagen Cross-linking Versus Epithelium-off Collagen Cross-linking in Pediatric Patients. Three Year Follow up.
Status: Completed | Type: Observational
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Luca Buzzonetti, Head of the Ophthalmology Department, Bambino Gesù IRCCS Children's Hospital, Rome, Italy, Bambino Gesù Hospital and Research Institute
Other Study IDs: PCXL
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iontophoretic transepithelial corneal cross-linking (I-ON CXL): Twenty eyes of 15 patients with keratoconus (mean age 13±3.5 [SD] years, range 9 to 18) underwent Iontophoresis epi-on CXL
  Interventions: Procedure: corneal cross-linking
- epithelium-off collagen cross-linking (epi-off CXL): Twenty eyes of 13 patients with keratoconus (14±4 [SD] years, range 10 to 18) underwent standard epi-off CXL
  Interventions: Procedure: corneal cross-linking

INTERVENTIONS:
Procedure: corneal cross-linking — Epithelium-off CXL was performed according to the Siena (Dresden modified) protocol: 2% pilocarpine was instilled 30 minutes before treatment, the epithelium was removed using a blunt knife. An isotonic solution of riboflavin 0.1% and dextran 20% was instilled for 10 minutes of corneal soaking before starting UV-A irradiation. The solution was administered every 3 minutes for a total of 30 minutes of UV-A exposure at 3mW/cm2.
  The iontophoresis device was filled with a hypoosmolar riboflavin 0.1% dextran-free solution enriched with ethylenediaminetetraacetic acid and trometamol. The device was then connected to a constant current generator initially set at 0.5 mA and increased to 1.0 mA to find out the individual tolerance. Iontophoresis was then performed for 5 minutes. The corneal device was then removed before performing UVA irradiation. During the irradiation phase (10 mW/cm2 for 9 minutes), good fluorescence was clearly detectable. The total treatment time was 14 minutes.

SUMMARY:
To compare 3 year iontophoretic transepithelial corneal cross-linking (I-ON CXL) outcomes with epithelium-off collagen cross-linking (epi-off CXL)in pediatric patients.

DETAILED DESCRIPTION:
Forty eyes of 28 consecutive pediatric patients (mean age 14.3±2.5 [SD] years; range, 9 to 18 years) with keratoconus were enrolled in the study. Twenty eyes of 15 patients underwent I-ON CXL, while 20 eyes of 13 patients underwent epi-off CXL. Corrected distance visual acuity (CDVA), spherical equivalent, maximum keratometry (Kmax), posterior elevation of the thinnest point and thickness of the thinnest point mean values were evaluated. A Student t test was used to compare baseline and 12, 24, and 36 month postoperative data. Keratoconus progression in function of preoperative Kmax value and cone location was evaluated at 36 months.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Keratoconus age < 18 years at the treatment; corneal cross linking performed at least 3 years before

Exclusion Criteria:

* age > 18 years at the treatment

Ages: 9 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Thirty eyes of 28 consecutive pediatric patients (7 female and 21 male; mean age 14.3±2.5 [SD] years; range, 9 to 18 years) affected by keratoconus (diagnosis established according to global consensus on keratoconus and ectatic diseases) who underwent iontophoresic transepithelial corneal cross-linking by or epithelium-off corneal cross-linking are enrolled in this retrospective study
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
keratoconus stability | 3 years
  To evaluate change of simulated maximum K (Kmax) that was calculated by a Sirius Scheimpflug camera (CSO, Firenze, Italy) by averaging the axial curvature from the fourth to the eighth Placido rings of the flattest and steepest meridians (the amplitude of the zone taken into consideration, therefore has a vari-able diameter depending on the curvature of the cornea, and the principal meridians are not nec-essarily 90 degrees away)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Buzzonetti, MD, Principal Investigator — Bambino Gesù Children's Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No